CLINICAL TRIAL: NCT05111509
Title: A Phase 0 First-in-human Clinical Trial of [203Pb]VMT-α-NET SPECT/CT for Somatostatin Receptor Imaging of Neuroendocrine Tumors
Brief Title: A First-in-human Clinical Trial to Evaluate an Alpha-radiation Imaging Agent
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yusuf Menda (Other)
Collaborators: Perspective Therapeutics (Industry); Holden Comprehensive Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Yusuf Menda, Professor and Director, Nuclear Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202006288; 5R01CA243014 (NIH)
Record Dates: First submitted 2021-10-30; First posted 2021-11-08 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Neuroendocrine Tumor Grade 2; Neuroendocrine Tumor Grade 1
Keywords: Alpha Particles; Pb-203 radioisotope; Single Photon Emission Computed Tomography Computed Tomography; SPECT CT Scan
MeSH Terms: interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- [203Pb]VMT-α-NET SPECT/CT (Experimental): injection of [203Pb]VMT-α-NET with serialized imaging and dosimetry measurements
  Interventions: Drug: [203Pb]VMT-α-NET; Device: SPECT/CT

INTERVENTIONS:
Drug: [203Pb]VMT-α-NET — 3 to 5 miliCuries of [203]Pb administered intravenously 60 minutes before the start of the scans.
Device: SPECT/CT — Scans are administered over 3 days: 1 hour post injection, 4 to 8 hours post-injection, 24 to 30 hours post-injection, and 42 to 52 hours post-injection.

SUMMARY:
This is a first in man study to determine if [203Pb]VMT-α-NET identifies neuroendocrine tumors with SPECT/CT. This is the first step to testing [212Pb]-based alpha radiation therapy in neuroendocrine therapy.

DETAILED DESCRIPTION:
The goal of this work is to use [203Pb]VMT-α-NET as the imaging agent to create a specialized patient treatment plan using [212Pb]VMT-α-NET as a first-in-human therapy for treatment resistant or refractory neuroendocrine tumors of the foregut or midgut. The first step is to test the imaging agent [203Pb]VMT-α-NET. This requires a very small dose of the drug (microdose) which is then measured by a series of images (like CT scans) over 4 days. Blood samples are also drawn that that time. It is hoped the imaging will identify the tumors so that a therapy using [212Pb]VMT-α-NET can be created.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to provide informed consent
* Stated willingness to comply with all study procedures and availability for duration of study
* Aged ≥ 18 years at the time of study drug administration
* Pathologically confirmed (histology or cytology) well-differentiated neuroendocrine tumor (WHO Grade 1 or 2) with primary location known or believed to be midgut or foregut
* At least 1 somatostatin receptor positive tumor site as demonstrated by PET/CT study utilizing an FDA approved PET agent within 12 months of consent
* ≥1 evaluable site of disease measuring ≥ 2.0 cm in any dimension on CT or MRI
* Adequate performance status (ECOG of 0 or 1; or KPS of ≥70).
* Not experiencing an uncontrolled intercurrent illness such as: infection requiring inpatient admission, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness/social situations, or any other condition that would limit compliance with study requirements as determined by study team members.

Exclusion Criteria:

* Individuals who are pregnant or breast feeding. A pregnancy test will be administered to individuals of child-bearing potential (per institutional policies) at screening. Individuals must agree to pregnancy tests prior to each administration of a radionuclidic agent for this study.
* Individuals of reproductive potential who decline to use effective contraception through the study (22 days equaling 10 half-lives).
* Lactating individuals who decline to withhold breastfeeding their child. As the effects of [203Pb]VMT-α-NET on the infant are unknown and relatively long half-life, women may not resume breast feeding for the current child.
* Therapeutic investigational drug within 4 weeks of C1D1
* Patients for whom, in the opinion of their physician, a 24-hour discontinuation of somatostatin analogue therapy represents a health risk.
* Subject's weight exceeds the limit of the imaging system.
* Long-acting somatostatin analogue treatment ≤ 20 days of C1D1
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to [90Y]DOTA-tyr3-Octreotide, Octreoscan®, or [68Ga]Octreotide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Ability of [203Pb]VMT-α-NET to identify neuroendocrine tumor lesions | Study days 1 through 5
  percentage of lesions detected with [203Pb]VMT-α-NET compared to the gold standard of NetSPOT or Ga-68 DOTATOC.

SECONDARY OUTCOMES:
Measure radiation dose from [203Pb]VMT-α-NET dosimetrically | Study days 1 through 5
  Determine the radiation absorbed dose to the organs and effective dose by pharmacokinetics through imaging and blood-measurements.
Single-time point survey | Study days 1 through 5
  Evaluate the potential of feasibility of single-time point imaging to measure the renal radiation dose

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Menda, M.D., Study Chair — University of Iowa
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared from those patient partners who agree to it. Data will be codified for the investigational team to provided additional details - as necessary - or confirm against source.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After study completion
Access Criteria: email the study chair; a non-disclosure and/or data usage agreement will most likely be required.